CLINICAL TRIAL: NCT00913926
Title: Multicenter Non-interventional Study on Efficacy, Tolerability, and Acceptance of Wellnara Containing 1.03 mg Estradiol Hemihydrate (Equivalent to 1 mg Estradiol) and 0.04 mg Levonorgestrel for Treatment of Hormone Deficiency Symptoms in Postmenopausal Women During 6 Cycles of 28 Days.
Brief Title: Effects of Wellnara on Climacteric Symptoms
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Jenapharm GmbH&Co.KG
Other Study IDs: 14575; WN0810DE (Other: Company Internal)
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Postmenopause
Keywords: Climacteric symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: E2/LNG oral (Wellnara, BAY86-5029)

INTERVENTIONS:
Drug: E2/LNG oral (Wellnara, BAY86-5029) — Patients in daily life treatment receiving Wellnara according to local drug information.

SUMMARY:
Aim of this NIS is to obtain further information on efficacy, tolerability, and acceptance of Wellnara in a large user population under the conditions of routine medical practice. Furthermore, any adverse drug reactions will be recorded in a large user population under the conditions of medical routine. To investigate the efficacy of Wellnara, patients will fill in a questionnaire, the so-called Menopause Rating Scale (MRS II). Further, the effects of treatment on skin and hair will be evaluated by the investigator. Patients will assess treatment effects on their sexual life. Safety parameters include monitoring of vaginal bleeding, measurement of blood pressure and body weight, and - as far as routinely used in the practice - calculation of waist-hip-ratio. Any relevant additional information related to adverse drug reactions will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* Women who have received a prescription of Wellnara on the basis of the decision of the treating gynecologist

Exclusion Criteria:

* Limited to the criteria listed in the expert information as contraindications

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study are women who have received a prescription of Wellnara on the basis of the decision of the treating gynecologist. The study is expected to collect data of up to 2,400 women in about 700 gynecological practices in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 749 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Primary endpoint in the observation of efficacy concerning climacteric complaints is the change in Menopause Rating Scale (MRS II) in relation to the status immediately before starting treatment (Baseline). | At Baseline, after 3 months, after 6 months

SECONDARY OUTCOMES:
Effects on climacteric-related skin, hair, and sexual problems | At Baseline, after 3 months, after 6 months
Subjective assessment of efficacy | After end of study
Body weight | At Baseline, after 3 months, after 6 months
Blood Pressure | At baseline, end of Study
Waist-hip-ratio (as far as routinely used in the practice) | At baseline, after 6 months
Occurrence of vaginal bleeding | After 3 months, after 6 months
Subjective assessment of tolerability | End of study
Adverse drug reactions | During the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany